CLINICAL TRIAL: NCT05732896
Title: Comparison of Opioid Consumption During Target Controlled Infusion (TCI) Guided by Nociception Level Index (NOL) or Standard Care Undergoing Intracranial Tumor Surgery, Randomized Controlled Study
Brief Title: Comparison of Opioid Consumption During TCI Guided by NOL Index or Standard Care Undergoing Intracranial Tumor Surgery
Acronym: NOLopioid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Turkish Society of Anesthesiology and Reanimation (Other)
Collaborators: Uludag University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: NOLguidedopioid
Record Dates: First submitted 2023-01-08; First posted 2023-02-17 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Target Controlled Infusion; Intracranial Neoplasm; Opioid; Nociceptive Pain; Anesthesia
Keywords: target controlled infusion; intraoperative nociception monitoring; Nociception Level index; neuroanesthesia; intracranial tumor surgery
MeSH Terms: conditions — Brain Neoplasms; Nociceptive Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): standard care group
- study group (Active Comparator): NOL guided group
  Interventions: Device: Nociception Leve Indeks

INTERVENTIONS:
Device: Nociception Leve Indeks — During TIVA-TCI, propofol (Schnider) effect site concentration (Ce) was titrated to BIS score between 40-60 and remifentanil (Minto) Ce to standard hemodynamic parameters in the control group and NOL index value between 10-25 in the study group.
  Arms: study group

SUMMARY:
In this prospective, randomized controlled study, we hypothesized that nociception level index monitoring reduced opioid administration during surgery. The secondary goals are to compare the total dose hypnotic drugs, as well as hemodynamic parameters, and to investigate the relationship between changes in the NOL index and HR change following severe noxious stimuli during effect site TCI of propofol and remifentanil in patients undergoing intracranial tumor surgery who are monitored using either standard monitors or the NOL monitor additionally.

DETAILED DESCRIPTION:
The study will be conducted on 50 patients aged between 18-75 years, with the American Society of Anesthesiologists (ASA) classification II-III, who would undergo intracranial tumor surgery after ethics committee approval (08/09/2020, 2020-15/15) and written consent from the patients. Standard monitoring (invasive arterial monitoring, 5-lead ECG, peripheral oxygen saturation-SpO2) and Bispectral Index Score (BIS) monitoring will be performed in the standard care group (SC; n=25), and NOL index monitoring will be performed in addition to standard monitors in the NOL guided group (NOL-G; n=25).

During TCI, propofol (Schnider) effect-site concentration (Ce) will be titrated to BIS score between 40-60 and remifentanil (Minto) Ce to standard hemodynamic parameters in the SC group and NOL index between 10-25 in the NOL-G group.

In all patients, Systolic, Diastolic and Mean Arterial Pressure (SAP, DAP, MAP), Heart Rate (HR), SpO2, BIS scores will be recorded before induction, intubation, head holder pinning, skin incision, muscle and periosteal dissection, craniotomy, dural incision, tumor excision, dural suturation, muscle and periosteum suturation, skin suturation, and interruption of infusions. In addition, NOL index in the NOL-G group patients will be recorded in all that time.

Hemodynamic parameters, to be administered propofol and remifentanil doses will be compared in two groups. NOL index changes before and after intubation, head holder pinning, skin incision and craniotomy, which are determined as severe noxious stimuli, will be compared with changes in HR.

Traditionally, the hemodynamic reactivity such as increased HR and blood pressure (BP), and/or nocifensive movements in the absence of paralytic agents are clinically considered for the assessment of nociception. The response to nociceptive stimuli is monitored as an increase in sympathetic or a decrease in parasympathetic tone (Guignard, 2006). The sympathetic response generates physiological changes such as increased HR, increased peripheral vasoconstriction, pupillary dilation, and changes in galvanic skin conductance (Guignard, 2006). As the understanding of nociception has grown in the past two decades, the industry has developed various nociception detecting devices based on some of the mentioned parameters.The only multi-parameter device is the Nociception Level (NOL) index (Ledowski, 2019). Evidence suggests the multi-parameter approach may be superior to the single-parameter approach for the assessment of nociceptive pain induced by tonic heat stimuli among healthy volunteers (Treister et al., 2012)

The PMD-200 system (NOL device) consists of a display and computing unit, a reusable non-invasive finger probe and a single-use sensor.The proprietary signal acquisition sensor platform (the combination of the finger probe and the single-use sensor) acquires physiological signals. Using advanced algorithms, the system processes and analyses multiple nociception related physiological parameters and their various derivatives, which correspond with the sympathetic nervous system's response to noxious stimuli. The finger probe and single-use sensor continuously acquire four physiological signals through the following four sensors; photoplethysmograph (PPG), galvanic Skin Response (GSR), peripheral Temperature (Temp), accelerometer (ACC). From these four signals the NOL algorithm extracts and analyses nociception-related physiological parameters and derivatives: pulse rate, pulse rate variability, pulse wave amplitude, skin conductance level, peripheral temperature, movement, and their various derivatives. Then a patient's specific nociception signature is established and continuously monitored. Peripheral temperature and movement serve as guardrails supporting algorithm validity and do not contribute directly to the algorithm calculation.

In 2013, Ben-Israel et al., published the first study on the multiparametric Nociception Level index (NOL). The few validation studies to date allowed the preliminary conclusion that the NOL index presented as an accurate means to measure the level of nociception during general anesthesia (Edry et al., 2016) . On the other hand, there are studies showing that the NOL index monitor does not reduce opioid consumption, or even though it does, there is no significant difference (Espitalier et al., 2021; F. Meijer et al., 2020; Niebhagen et al., 2022; Renaud-Roy et al., 2022) In addition, many studies in the literature indicate that NOL index monitoring is a reliable monitor in the evaluation of nociception or in distinguishing noxius stimuli (Renaud-Roy et al., 2019) (Treister et al., 2012) (Edry et al., 2016) (Martini et al., 2015) (Bollag et al., 2018) .

ELIGIBILITY:
Inclusion Criteria:

* İntracranial mass surgery
* Craniotomy
* ASA II-II
* elective surgery

Exclusion Criteria:

* pregnant or suspected of pregnancy
* receive antiarrhythmic therapy
* autonomic nervous system disease
* ASA IV
* emergency surgery
* patients with difficult airway features
* patients receiving chronic pain treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
comparison of administered remifentanil doses (mcg/kg/min) | throughout the operation
  This data will be obtained from the TCI device. Demographic data such as the patient's gender, age, weight, etc. are entered into the TCI device. The TCI device displays the total duration of the operation as hour and the total amount of drug used as microgram.
  To control for patient weight and duration of surgery, we report the anesthesia drug doses as dose/kg/min of anesthesia time.The remifentanil administration dose is indicated in mcg/kg/min.
  "kg" is patient's actual body weight. "min" is operating time in minutes.

SECONDARY OUTCOMES:
comparison of hemodynamic parameters | throughout the operation
  Standard (invasive arterial monitoring, 5-lead ECG, peripheral oxygen saturation-SpO2) and BIS monitoring will be performed in the SC group, and NOL index monitoring will be performed in addition to standart monitors in the NOL-G group.
  SAP, DAP, MAP, HR will be recorded before induction (T0), intubation (T1), head holder pinning (T2), skin incision (T3), muscle and periosteal dissection (T4), craniotomy (T5), dural incision (T6), tumor excision (T7), dural suturation (T8), muscle and periosteum suturation(T9), skin suturation (T10), and interruption of infusions (T11).
  Hemodynamic parameters and BIS score are recorded on the anesthesia device monitor.
  SAP, DAP, MAP are defined as mmhg. HR is defined as beat per minute BIS score and NOL index give an index between 0-100. NOL index device saves data itself and this data can be exported via flash memory.
comparison of variability NOL index during severe noxious stimuli | throughout the operation
  NOL index changes before and after intubation, head holder pinning, skin incision, and craniotomy, which were determined and compared as severe noxious stimuli.
  The NOL index device records the heart rate and the NOL index every 5 seconds.
comparison of variability Heart rate during severe noxious stimuli | throughout the operation
  Heart rate changes before and after intubation, head holder pinning, skin incision, and craniotomy, which were determined and compared as severe noxious stimuli.
  The NOL index device records the heart rate and the NOL index every 5 seconds.
comparison of administered propofol dose (mg/kg/min) | throughout the operation
  This data will be obtained from the TCI device. Demographic data such as the patient's gender, age, weight, etc. are entered into the TCI device. The TCI device displays the total duration of the operation as hour and the total amount of drug used as milligram.
  To control for patient weight and duration of surgery, we report the anesthesia drug doses as dose/kg/min of anesthesia time. The propofol administration dose is indicated in mg/kg/min.
  "kg" is patient's actual body weight. "min" is operating time in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Hulya Bilgin, Study Director — Bursa Uludağ University Faculty of Medicine Department of Anesthesiology and Reanimation
Locations (1):
- Uludag University Medical Faculty, Bursa, Nilufer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guignard B. Monitoring analgesia. Best Pract Res Clin Anaesthesiol. 2006 Mar;20(1):161-80. doi: 10.1016/j.bpa.2005.09.002. PMID 16634423
- [Background] Ledowski T. Objective monitoring of nociception: a review of current commercial solutions. Br J Anaesth. 2019 Aug;123(2):e312-e321. doi: 10.1016/j.bja.2019.03.024. Epub 2019 Apr 30. PMID 31047645
- [Result] Ben-Israel N, Kliger M, Zuckerman G, Katz Y, Edry R. Monitoring the nociception level: a multi-parameter approach. J Clin Monit Comput. 2013 Dec;27(6):659-68. doi: 10.1007/s10877-013-9487-9. Epub 2013 Jul 9. PMID 23835792
- [Result] Edry R, Recea V, Dikust Y, Sessler DI. Preliminary Intraoperative Validation of the Nociception Level Index: A Noninvasive Nociception Monitor. Anesthesiology. 2016 Jul;125(1):193-203. doi: 10.1097/ALN.0000000000001130. PMID 27171828
- [Result] Funcke S, Pinnschmidt HO, Brinkmann C, Wesseler S, Beyer B, Fischer M, Nitzschke R. Nociception level-guided opioid administration in radical retropubic prostatectomy: a randomised controlled trial. Br J Anaesth. 2021 Feb;126(2):516-524. doi: 10.1016/j.bja.2020.09.051. Epub 2020 Nov 20. PMID 33228979
- [Result] Ma D, Ma J, Chen H, Mu D, Kong H, Yu L. Nociception monitors vs. standard practice for titration of opioid administration in general anesthesia: A meta-analysis of randomized controlled trials. Front Med (Lausanne). 2022 Aug 25;9:963185. doi: 10.3389/fmed.2022.963185. eCollection 2022. PMID 36091708
- [Result] Meijer FS, Martini CH, Broens S, Boon M, Niesters M, Aarts L, Olofsen E, van Velzen M, Dahan A. Nociception-guided versus Standard Care during Remifentanil-Propofol Anesthesia: A Randomized Controlled Trial. Anesthesiology. 2019 May;130(5):745-755. doi: 10.1097/ALN.0000000000002634. PMID 30829658
- [Result] Espitalier F, Idrissi M, Fortier A, Belanger ME, Carrara L, Dakhlallah S, Rivard C, Brulotte V, Zaphiratos V, Loubert C, Godin N, Fortier LP, Verdonck O, Richebe P. "Impact of Nociception Level (NOL) index intraoperative guidance of fentanyl administration on opioid consumption, postoperative pain scores and recovery in patients undergoing gynecological laparoscopic surgery. A randomized controlled trial". J Clin Anesth. 2021 Dec;75:110497. doi: 10.1016/j.jclinane.2021.110497. Epub 2021 Sep 28. PMID 34597955
- [Result] Meijer F, Honing M, Roor T, Toet S, Calis P, Olofsen E, Martini C, van Velzen M, Aarts L, Niesters M, Boon M, Dahan A. Reduced postoperative pain using Nociception Level-guided fentanyl dosing during sevoflurane anaesthesia: a randomised controlled trial. Br J Anaesth. 2020 Dec;125(6):1070-1078. doi: 10.1016/j.bja.2020.07.057. Epub 2020 Sep 17. PMID 32950246
- [Result] Niebhagen F, Golde C, Koch T, Hubler M. [Does NoL monitoring affect opioid consumption during da Vinci prostatectomy?]. Anaesthesiologie. 2022 Sep;71(9):683-688. doi: 10.1007/s00101-022-01126-7. Epub 2022 May 25. German. PMID 35925157
- [Result] Renaud-Roy E, Morisson L, Brulotte V, Idrissi M, Godin N, Fortier LP, Verdonck O, Choiniere M, Richebe P. Effect of combined intraoperative use of the Nociception Level (NOL) and bispectral (BIS) indexes on desflurane administration. Anaesth Crit Care Pain Med. 2022 Jun;41(3):101081. doi: 10.1016/j.accpm.2022.101081. Epub 2022 Apr 25. PMID 35472586
- [Result] Renaud-Roy E, Stockle PA, Maximos S, Brulotte V, Sideris L, Dube P, Drolet P, Tanoubi I, Issa R, Verdonck O, Fortier LP, Richebe P. Correlation between incremental remifentanil doses and the Nociception Level (NOL) index response after intraoperative noxious stimuli. Can J Anaesth. 2019 Sep;66(9):1049-1061. doi: 10.1007/s12630-019-01372-1. Epub 2019 Apr 17. PMID 30997633
- [Result] Treister R, Kliger M, Zuckerman G, Aryeh IG, Eisenberg E. Differentiating between heat pain intensities: the combined effect of multiple autonomic parameters. Pain. 2012 Sep;153(9):1807-1814. doi: 10.1016/j.pain.2012.04.008. Epub 2012 May 29. PMID 22647429
- [Result] Martini CH, Boon M, Broens SJ, Hekkelman EF, Oudhoff LA, Buddeke AW, Dahan A. Ability of the nociception level, a multiparameter composite of autonomic signals, to detect noxious stimuli during propofol-remifentanil anesthesia. Anesthesiology. 2015 Sep;123(3):524-34. doi: 10.1097/ALN.0000000000000757. PMID 26154185